CLINICAL TRIAL: NCT05358249
Title: KontRASt-03: A Phase Ib/II, Multicenter, Open-label Platform Study of JDQ443 With Select Combinations in Patients With Advanced Solid Tumors Harboring the KRAS G12C Mutation
Brief Title: Platform Study of JDQ443 in Combinations in Patients With Advanced Solid Tumors Harboring the KRAS G12C Mutation
Acronym: KontRASt-03
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJDQ443E12101; 2021-006196-42 (EudraCT Number)
Expanded Access: NCT05038631 (Available)
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: KRAS G12C Mutant Solid Tumors; Carcinoma, Non-Small Cell Lung; Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Colorectal Cancer; Colorectal Carcinoma; Colorectal Neoplasms; Colorectal Tumors; Neoplasms, Colorectal
Keywords: KRAS G12C; targeted therapy; NSCLC; CRC; advanced solid tumors; JDQ443; trametinib; ribociclib; cetuximab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — JDQ443; trametinib; ribociclib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JDQ443+trametinib (Experimental): JDQ443 in combination with trametinib
  Interventions: Drug: JDQ443; Drug: trametinib
- JDQ443+ribociclib (Experimental): JDQ443 in combination with ribociclib
  Interventions: Drug: JDQ443; Drug: Ribociclib
- JDQ443+cetuximab (Experimental): JDQ443 in combination with cetuximab
  Interventions: Drug: JDQ443; Biological: cetuximab

INTERVENTIONS:
Drug: JDQ443 — KRAS G12C inhibitor, oral
Drug: trametinib — MEK inhibitor, oral
  Other Names: TMT212
  Arms: JDQ443+trametinib
Drug: Ribociclib — CDK4/6 inhibitor, oral
  Other Names: LEE011
  Arms: JDQ443+ribociclib
Biological: cetuximab — EGFR inhibitor, intravenous
  Arms: JDQ443+cetuximab

SUMMARY:
This is Phase Ib/II, multicenter, open-label adaptive platform study of JDQ443 with select therapies in patients with advanced solid tumors harboring the KRAS G12C mutation.

DETAILED DESCRIPTION:
JDQ443 will be considered "backbone" treatment in this trial and combined with selected therapies, or "partner(s)". The combination of a backbone and a partner will constitute a treatment arm. After dose escalation, treatment arms that reach a maximum tolerated dose /recommended dose and are determined to be safe may, but are not required to, proceed to Phase II to further explore safety, tolerability, and anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation:

- Patients with advanced (metastatic or unresectable) KRAS G12C mutant solid tumors who have received standard of care therapy or are ineligible to receive such therapy.

Phase II:

* Patients with advanced (metastatic or unresectable) KRAS G12C mutant non-small cell lung cancer who have received platinum-based chemotherapy regimen and immune checkpoint inhibitor therapy, unless patient was ineligible to receive such therapy
* Patients with advanced (metastatic or unresectable) KRAS G12C mutant colorectal cancer who have received fluropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, unless patient was ineligible to such therapy.

All patients:

* ECOG performance status of 0 or 1.
* Patients must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines.

Exclusion Criteria:

* Tumors harboring driver mutations that have approved targeted therapies, with the exception of KRAS G12C mutations
* Prior treatment with a KRAS G12C inhibitor is excluded for patients in a subset of groups in Phase II.
* Active brain metastases, including symptomatic brain metastases or known leptomeningeal disease
* Clinically significant cardiac disease or risk factors at screening
* Insufficient bone marrow, hepatic or renal function at screening Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Incidence and severity of dose limiting toxicities (DLTs) of each combination treatment. | 28 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value that is not primarily related to disease, disease progression, intercurrent illness/injury, or concomitant medications that occurs within the first 28 days of study treatment and meets a defined criteria.
Dose escalation: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) by treatment | 24 months
  All information obtained on AE will be displayed by treatment group. Summary tables will include only AEs that started/worsened during the cycles of treatment (treatment-emergent AEs).
Dose escalation: Frequency of dose interruptions and reductions, by treatment | 24 months
  The number of patients with dose adjustments (reductions and interruptions) will be summarized by treatment group.
Dose Escalation: Dose intensity by treatment | 24 months
  Dose intensity is defined as the ratio of actual cumulative dose received and actual duration of response.
PhaseII: Overall Response Rate by Blinded Independent Review Committee (BIRC) per RECIST 1.1 | 24 months
  ORR is the proportion of patients with a best overall response (BOR) of Complete Response (CR) or Partial Response (PR).

SECONDARY OUTCOMES:
Dose escalation and Phase II: ORR by local review per RECIST 1.1 | 24 months
  ORR is the proportion of patients with a BOR of CR or PR.
Dose escalation and Phase II: Disease Control Rate (DCR) by local review per RECIST 1.1 | 24 months
  DCR is the proportion of patients with a BOR of CR or PR or Stable Disease (SD). The objective of this endpoint is to summarize patients with signs of "activity" defined as either shrinkage of tumor (regardless of duration) or slowing down of tumor growth.
Dose escalation and Phase II: Duration of Response (DoR) by local review per RECIST 1.1 | 24 months
  Duration of response is defined as the time from the date of the first documented response (CR or PR), to the date of first documented progression, or death due any cause.
Dose escalation and Phase II: Progression-Free Survival (PFS) by local review per RECIST 1.1 | 24 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression, or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Phase II: DCR by BIRC per RECIST 1.1 | 24 months
  DCR is the proportion of patients with a BOR of CR or PR or SD. The objective of this endpoint is to summarize patients with signs of "activity" defined as either shrinkage of tumor (regardless of duration) or slowing down of tumor growth.
Phase II: DoR by BIRC per RECIST 1.1 | 24 months
  Duration of response is defined as the time from the date of the first documented response (CR or PR), to the date of first documented progression, or death due any cause.
Phase II: PFS by BIRC per RECIST 1.1 | 24 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression, or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Phase II: Overall survival (OS) | 24 months
  OS is defined as the time from date of randomization/start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last known date patient alive.
Dose escalation and Phase II: PK parameters - Maximum Concentration (Cmax), as applicable per arm | 5 months
  The maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass x volume-1)
Dose escalation and Phase II: PK parameters - Minimum Concentration (Cmin), as applicable per arm | 5 months
  Observed concentration at the end of a dosing interval (taken directly before next administration)
Dose escalation: Time to achieve Cmax - Tmax, as applicable per arm | 5 months
  The time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (time)
Dose escalation and Phase II: Plasma or serum concentration vs time profiles - AUCtau, as applicable per arm | 5 months
  The Area under curve calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1)
Dose escalation and Phase II: Plasma or serum concentration vs time profiles - AUCinf, as applicable per arm | 5 months
  The AUC from time zero to infinity (mass x time x volume-1)
Phase II: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) by treatment | 24 months
  All information obtained on AE will be displayed by treatment group. Summary tables will include only AEs that started/worsened during the cycles of treatment (treatment-emergent AEs).
Phase II: Frequency of dose interruptions and reductions, by treatment | 24 months
  The number of patients with dose adjustments (reductions and interruptions) will be summarized by treatment group.
Phase II: Dose intensity by treatment | 24 months
  Dose intensity is defined as the ratio of actual cumulative dose received and actual duration of response.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYU School of Medicine, New York, New York
- Novartis Investigative Site, Leuven, Belgium
- France (2):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
- Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.